CLINICAL TRIAL: NCT02562794
Title: Addressing Mental Health Disparities in Refugee Children: A CBPR Collaboration
Brief Title: Addressing Mental Health Disparities in Refugee Children: A Community-based Participatory Research (CBPR) Collaboration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Theresa Betancourt, Salem Professor in Global Practice, Boston College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15860; R24MD008057 (NIH)
Record Dates: First submitted 2015-07-22; First posted 2015-09-29 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Child/Adolescent Problems; Mental Disorders
Keywords: refugee
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Family Strengthening Intervention-Refugees. A total of 20 Somali Bantu and 20 Bhutanese refugee families will participate in a Family Strengthening Intervention adapted for use with refugees.
  Interventions: Behavioral: Family Strengthening Intervention-Refugees
- Control (No Intervention): A total of 20 Somali Bantu and 20 Bhutanese refugee families will receive services as usual.

INTERVENTIONS:
Behavioral: Family Strengthening Intervention-Refugees — This study aims to design a preventive intervention for at-risk refugee children and families. The intervention is focused on strengthening core family resources and promoting resilience and healthy parent-child interactions.
  Arms: Intervention

SUMMARY:
This study will use CBPR mixed methods (qualitative and quantitative data collection) to conduct needs assessments and design and evaluate a core family-based intervention. Project activities will emphasize capacity building in two refugee communities resettled in Greater Boston-the Somali Bantu and the Bhutanese-actively engaging refugee community members, community advisory boards, services providers, and other stakeholders. Specific Aims are to: (1) deepen partnerships with the Somali Bantu and Bhutanese communities through co-leadership, capacity-building, and knowledge sharing; (2) collect and apply qualitative data to (a) prepare a needs assessment of mental health in children and adolescents, barriers to care, and services preferences with each target refugee group; (b) develop mental health/psychosocial assessments for refugee caregivers and children; (c) adapt the core components of a family-based strengthening intervention for use with refugees; and (3) conduct an 80-family pilot study to examine acceptability and sustainability of the intervention. Key outcomes will be reduced mental health symptoms among children and adolescents and improvement in caregiver-child relationships.

DETAILED DESCRIPTION:
The proposed mixed methods study will apply CBPR methods in an innovative, cross-cultural project to assess mental health problems in children and community strengths in two refugee communities-the Somali Bantu and the Bhutanese-and to design and pilot test a family-based intervention for refugees in their native languages (Somali Bantu Maay Maay and the Nepali language used by Bhutanese refugees). We will use qualitative research methods developed in preliminary research with the Somali Bantu to identify local conceptualizations of mental health problems, resilience, attitudes about healing and help-seeking, and preferences for mental health services among resettled Bhutanese. The CBPR team will collaborate on mental health needs assessments for both communities, with attention paid to shared experiences and strengths.

Findings on risk and protective factors influencing child mental health will inform development of a preventive intervention. Community Advisory Boards (CABs) will actively participate in the review and selection of intervention components. Based on preliminary research with the Somali Bantu community, we anticipate that a family-based intervention model will respond well to community requests for parenting support and psychoeducation about trauma and effects in families. An intervention positively oriented towards existing sources of family resilience and self-efficacy has great potential for improving access to and engagement in mental health care and other social services, and for increasing both formal and non-formal supports-all essential for reducing mental health disparities.

In this manner, community and university partners will collaborate to achieve four Specific Aims:

Aim 1: Strengthen existing relationships and decision-making partnerships with the Somali Bantu and Bhutanese refugee communities in Greater Boston through community based participatory research in partnership with the Shanbaro Community Association and Chelsea Collaborative in Chelsea, Massachusetts.

Aim 2: Collect and analyze qualitative data on local conceptualizations of mental health problems and resilience in school-age children (ages 5-17) as well as help seeking and services preferences among Somali Bantu and Bhutanese refugee families; use findings to inform intervention targets and critical components of a family-based preventive intervention, the Family Strengthening Intervention (FSI) for refugees.

Aim 3: Use qualitative findings to prepare (a) a needs assessment of mental health in school-age children, community strengths, barriers to care, and services preferences with each target refugee group; (b) a preliminary battery of mental health/psychosocial measures for use in mental health assessment of children and caregivers; and (c) a draft set of intervention, recruitment, and training materials.

Aim 4: Use CBPR approaches to recruit and enroll 80 families in a feasibility study, with half randomized to care as usual and half to the FSI delivered by trained community interventionists; conduct longitudinal assessments at baseline, post-intervention, and 6 months. Hypothesis 4.1: Participation in the refugee FSI will be associated with improved communication and connectedness within families, increased mental health services access, and increased knowledge among caregivers and children on the consequences of trauma in refugee families. Hypothesis 4.2: Participation in the refugee FSI will be associated with increased application of healthy parenting skills, parental self-efficacy, parental supervision of children, improved functioning and reduced symptoms of internalizing and externalizing in school-age refugee children.

ELIGIBILITY:
Inclusion Criteria:

* Refugee families must have a school-aged child (aged 5-17), and caregivers must be at least 18 years of age and live in the same household as the child.

Exclusion Criteria:

* Untreated mental illness or active family crisis

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms among children and adolescents | Depressive symptoms will be measured at three time points - at baseline prior to intervention, immediately post-intervention (an average of 16 weeks after baseline), and 6 months after the completion of the intervention
  Depressive symptoms will be measured with an adapted version of the Center for Epidemiologic Study-Depression) CES-D scale

SECONDARY OUTCOMES:
Change in anxiety symptoms among children and adolescents | Anxiety symptoms will be measured at three time points - at baseline prior to intervention, immediately post intervention (an average of 16 weeks after baseline), and six months after the completion of the intervention
  Anxiety symptoms will be measured with an adapted version of the CES-D
Change in externalizing/behavioral problems among children and adolescents | Externalizing symptoms will be measured at three time points - at baseline prior to intervention, immediately post-intervention (an average of 16 weeks after the baseline), and 6 months after the completion of the intervention
  Externalizing symptoms will be measured with the (Youth Self-Report) YSR externalizing sub scale
Change in parent-child relationships | Quality of parent-child relationships will be measured at three time points - at baseline prior to intervention, immediately post-intervention (an average of 16 weeks after the baseline), and 6 months after the completion of the intervention.
  Parent-child relationships will be measured with an adapted version of the Alabama parenting scale

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Betancourt, ScD, Principal Investigator — Boston College
Locations (2):
- United States (2):
  - Chelsea Collaborative, Chelsea, Massachusetts
  - Jewish Family Service, Springfield, Massachusetts

REFERENCES:
- [Background] Betancourt TS, Frounfelker R, Mishra T, Hussein A & Falzarano R. American Journal of Public Health. Published on-line ahead of print April 23, 2015; e1-8. doi:10.2105/AJPH.2014.302504